CLINICAL TRIAL: NCT02004288
Title: The Role of Lactobacillus Reuteri in Nutritional Recovery and Treatment of Constipation in Children and Adolescents With Anorexia Nervosa - Randomised, Double Blind, Placebo Controlled Study
Brief Title: The Role of Lactobacillus Reuteri in Children and Adolescents With Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CSUB0083
Record Dates: First submitted 2013-12-02; First posted 2013-12-09 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-05

CONDITIONS: Anorexia Nervosa; Constipation
Keywords: Probiotics; Anorexia nervosa; Constipation; Body weight
MeSH Terms: conditions — Anorexia Nervosa; Constipation; Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus reuteri Protectis DSM17938 (Experimental): One chewable tablet twice per day with L reuteri Protectis DSM 17938, 1x108 CFU/tablet (colony forming unit)
  Interventions: Dietary Supplement: Lactobacillus reuteri Protectis DSM17938
- Placebo (Placebo Comparator): One chewable tablet twice per day with placebo per day
  Interventions: Dietary Supplement: Lactobacillus reuteri Protectis DSM17938

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri Protectis DSM17938 — One chewable tablet with L. reuteri or placebo taken twice a day for 3 months. After the 3 month therapy both groups will be monitored for the next 3 months.

SUMMARY:
The aim of this study is to investigate whether Lactobacillus reuteri could have a beneficial role in treatment of children and adolescents with Anorexia nervosa who develop motility disorder due to the malnutrition regarding the normalization of the motility, as well as the possible role of probiotics on nutritional recovery, especially on bone health.

DETAILED DESCRIPTION:
Pediatric patients with AN and constipation referred to gastroenterologist for nutritional rehabilitation at the Department of Pediatric Gastroenterology, Hepatology and Nutrition, Clinical Hospital Center Sestre Milosrdnice, Zagreb, approximately 30 children, will be asked to participate.

The evaluation of patients will be conducted through APA DSM-V diagnostic criteria for anorexia nervosa and Rome III criteria for constipation.

During the hospitalization all of the patients will receive conventional nutritional rehabilitation that is composed of serving normal food under supervision of nurses that calculate daily caloric intake through 5-6 meals and according to that additional enteral nutrition that consist of polymeric enteral formula. Daily caloric intake is calculated as kcal/kg/day and is slowly rising through 2 weeks starting from 80% to the goal of 130% of daily energy requirements according to FAO 2004 recommendation.

Anthropometry measures will be taken at the time of hospitalization and at every visit.

Normalization of weight is when the Z-score for BMI is less than -1.5 according to CDC BMI-growth charts, or normalisation of menstrual cycle is achieved.

In order to achieve adherence to therapeutic protocol parents will be contacted by phone at least once in 7-10 days. Participants will be instructed to keep diary on a daily basis (adherence to therapy, stool diary). All patients will return packages with all used, and unused product.

BASELINE -VISIT 1 Randomization at first day of hospitalization. In all patients anthropometry will be performed at the time of hospitalization, as well as dual-energy X-ray absorptiometry (DEXA) and serum D3 levels at first 2 days of hospitalization as a part of routine diagnostic protocol in heavily underweight patients with AN.

VISIT 2 4 weeks after randomization, at discharge from hospital Anthropometry

VISIT 3 8 weeks after randomization, 4 weeks after discharge from hospital Anthropometry

END OF STUDY -VISIT 4 3 months after baseline Anthropometry

VISIT 5 3 months after the end of study (6 months after baseline) At this point control serum D3 levels and DEXA will be performed at all patients Anthropometry

All the symptoms and daily caloric intake will be monitored using diaries attached to protocol.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with Anorexia nervosa and constipation, aged 8-18 years

Exclusion Criteria:

* AN and constipation present for less than 3 month prior to hospitalization
* any disease that affects GI or other systems other than AN or functional constipation
* chronic disorder other than AN
* receiving probiotic and/or prebiotic products 14 days prior to enrolment
* receiving antibiotics 14 days prior to enrolment
* constipation prior AN
* receiving laxative as a therapy for constipation or abuse of laxative to lose weight prior to enrolment
* extraintestinal symptoms: fever, rash
* abnormalities in laboratory findings
* abnormalities in clinical findings: organomegaly, perianal disease

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2013-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orjena Zaja Franulovic, MD, PhD, Principal Investigator — Center for Eating disorders Sestre milosrdnice University hospital Zagreb, Croatia
Locations (1):
- Pediatric Department Clinical Hospital Centre Sestre milosrdnice Gastroenterology, Hepatology and Nutrition Ward, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zaja O, Fiolic M, Cuk MC, Tiljak MK. "The role of L. reuteri DSM17938 in nutritional recovery and treatment of constipation in children and adolescents with anorexia nervosa - a randomized, double blind, placebo controlled study". Clin Nutr ESPEN. 2021 Dec;46:47-53. doi: 10.1016/j.clnesp.2021.08.016. Epub 2021 Sep 8. PMID 34857236

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lactobacillus Reuteri Protectis DSM17938 | Placebo
Started | 15 | 16
Completed | 14 | 15
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactobacillus Reuteri Protectis DSM17938 | Placebo | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 16 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.06 (2.31) | 15.13 (1.70) | 15.06 (1.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Croatia | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Drop Out From Rome III Criteria for Constipation
Description: Drop out from Rome III criteria for constipation: Yes / No. According to Rome III, a diagnosis of functional constipation is made when at least two of the following criteria are met for the last 3 months with symptom onset at least 6 months prior to diagnosis: a) straining on >25% of defecations; b) lumpy or hard stools on >25% of defecations; c) sensation of incomplete evacuation on >25% of defecations; d) sensation of anorectal obstruction/blockage on >25% of defecations; e) manual maneuvers on >25% of defecations; and f) less than 3 defecations per week.
Time Frame: 3 month
Measure: Count of Participants; unit: Participants
Arm/Group | Lactobacillus Reuteri Protectis DSM17938 | Placebo
Number analyzed (Participants) | 15 | 16
Participants | 13 | 10

2. Secondary Outcome: Normalization of Body Weight
Description: normalization of body weight- 90% of premorbid weight, or ≥10. centile for BMI (according to the WHO growth charts)
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Lactobacillus Reuteri Protectis DSM17938 | Placebo
Number analyzed (Participants) | 15 | 16
Participants | 14 | 10

ADVERSE EVENTS:
Time Frame: During the study, 6 months / participant,
Arm/Group | Lactobacillus Reuteri Protectis DSM17938 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

LIMITATIONS AND CAVEATS:
The limitation of this study is the small number of patients. This is due to strict inclusion and exclusion criteria, as well as the fact that some parents and patients refused to participate in the survey, which is not unusual given the negativism that characterizes this disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No